CLINICAL TRIAL: NCT04857034
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of Deucravacitinib (BMS-986165) in Participants With Active Discoid and/or Subacute Cutaneous Lupus Erythematosus (DLE/SCLE)
Brief Title: A Study to Evaluate Efficacy and Safety of Deucravacitinib in Participants With Active Discoid and/or Subacute Cutaneous Lupus Erythematosus (DLE/SCLE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-132; 2020-000071-21 (EudraCT Number); U1111-1246-1726 (Registry Identifier: WHO)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Lupus Erythematosus, Discoid; Lupus Erythematosus, Subacute Cutaneous
Keywords: BMS-986165; Deucravacitinib; DLE; Discoid Lupus Erythematosus; SCLE; Subacute Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid; Lupus Erythematosus, Cutaneous | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Treatment: Deucravacitinib Dose 1 (Experimental)
  Interventions: Drug: Deucravacitinib
- Active Treatment: Deucravacitinib Dose 2 (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Arms: Active Treatment: Deucravacitinib Dose 1; Active Treatment: Deucravacitinib Dose 2
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, efficacy, and tolerability of deucravacitinib (BMS-986165) compared with placebo in participants with active discoid and/or subacute cutaneous lupus erythematosus (DLE/SCLE). This study will also assess if deucravacitinib is biologically active and potentially effective in the treatment of participants with moderate to severe DLE/SCLE with or without systemic lupus erythematosus (SLE) that is not well controlled with standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of discoid/subacute cutaneous lupus erythematosus (DLE/SCLE) for at least 3 months prior to screening visit
* Meets both clinical and histopathological diagnostic cutaneous lupus erythematosus (CLE) criteria per protocol
* Currently receiving treatment for DLE/SCLE with a stable regimen of at least one of the following medications: oral corticosteroid, and/or antimalarial, and/or immunosuppressant
* Participant could be with or without concurrent systemic lupus erythematosus (SLE)
* If participant receives nonsteroidal anti-inflammatory drugs (NSAIDs) or analgesics treatment then the participant must be on a stable dose 2 weeks prior to screening

Exclusion Criteria:

* Women who are pregnant, lactating, breastfeeding or planning pregnancy during the study period
* Any of the following specific CLE subtypes in isolation: acute cutaneous lupus erythematosus (ACLE), lupus tumidus, lupus (profundus) panniculitis, chilblains
* Drug-induced CLE and/or drug-induced systemic lupus erythematosus (SLE)
* Antiphospholipid antibody syndrome, serious thrombotic event or unexplained pregnancy loss within 1 year before the screening visit
* History of 3 or more unexplained consecutive pregnancy losses
* Active severe or unstable neuropsychiatric SLE
* Other autoimmune diseases or non-SLE driven inflammatory joint or skin disease or overlap syndromes as primary disease that in the opinion of the investigator will significantly impact the assessment of CLE/SLE disease manifestations and activity

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2028-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (41):
- United States (12):
  - Local Institution - 0077, Scottsdale, Arizona
  - Local Institution - 0076, Irvine, California
  - Local Institution - 0046, Los Angeles, California
  - Local Institution - 0073, Farmington, Connecticut
  - Local Institution - 0082, Orlando, Florida
  - Local Institution - 0060, Ann Arbor, Michigan
  - Local Institution - 0059, St Louis, Missouri
  - Local Institution - 0037, New York, New York
  - Local Institution - 0065, Durham, North Carolina
  - Local Institution - 0067, Columbus, Ohio
  - Local Institution - 0026, Oklahoma City, Oklahoma
  - Local Institution - 0054, Charleston, South Carolina
- Argentina (3):
  - Local Institution - 0018, Capital Federal, Buenos Aires
  - Local Institution - 0013, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0019, Buenos Aires
- Australia (6):
  - Local Institution - 0003, Botany, New South Wales
  - Local Institution - 0001, Kogarah, New South Wales
  - Local Institution - 0002, Camberwell, Victoria
  - Local Institution - 0007, Clayton, Victoria
  - Local Institution - 0078, Melbourne, Victoria
  - Local Institution - 0087, Victoria Park, Western Australia
- France (3):
  - Local Institution - 0038, Bordeaux
  - Local Institution - 0027, Créteil
  - Local Institution - 0010, Paris
- Germany (4):
  - Local Institution - 0072, Dresden, Saxony
  - Local Institution - 0035, Berlin
  - Local Institution - 0014, Erlangen
  - Local Institution - 0006, Hamburg
- Mexico (6):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution - 0058, Zapopan, Jalisco
  - Local Institution - 0036, Monterrey, Nuevo León
  - Local Institution - 0029, Aguascalientes
  - Local Institution - 0028, Guadalajara
  - Local Institution - 0071, Mexico City
- Poland (3):
  - Local Institution - 0005, Rzeszów
  - Local Institution - 0009, Wroclaw
  - Local Institution - 0008, Lodz, Łódź Voivodeship
- Taiwan (4):
  - Local Institution - 0031, Kaohsiung City
  - Local Institution - 0023, Taichung
  - Local Institution - 0021, Taichung
  - Local Institution - 0022, Taipei

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04857034.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 participants randomized and 73 treated in the placebo controlled period. 18 participants who received placebo in the placebo controlled period were randomized into 2 separate treatment arms during active treatment period.
Groups:
- Placebo-Controlled Period: Treatment 1: Deucravactinib 3mg
- Placebo-Controlled Period: Treatment 2: Received Deucravacitinib 6mg in placebo controlled period and Deucravacitinib 6mg in active treatment period
- Placebo-Controlled Period: Placebo: Placebo
- Active-Treatment Period: Treatment 1: Deucravacitinib 3mg
- Active-Treatment Period: Treatment 2: Deucravacitinib 6mg
Period: Placebo-Controlled Period
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo | Active-Treatment Period: Treatment 1 | Active-Treatment Period: Treatment 2
Started (= randomized) | 25 | 25 | 24 | 0 | 0
Completed | 21 | 20 | 22 | 0 | 0
Not Completed | 4 | 5 | 2 | 0 | 0
Not completed — Request to discontinue | 2 | 2 | 0 | 0 | 0
Not completed — withdrew consent | 1 | 1 | 2 | 0 | 0
Not completed — Pregnancy | 1 | 1 | 0 | 0 | 0
Not completed — Ongoing study period | 0 | 1 | 0 | 0 | 0
Period: Active Treatment Period
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo | Active-Treatment Period: Treatment 1 | Active-Treatment Period: Treatment 2
Started (= started treatment in acitive treatment period) | 16 | 20 | 0 | 9 | 9
Completed | 11 | 9 | 0 | 5 | 6
Not Completed | 5 | 11 | 0 | 4 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — request to discontinue | 0 | 1 | 0 | 1 | 0
Not completed — administrative reason by sponsor | 1 | 5 | 0 | 2 | 2
Not completed — other reasons | 1 | 1 | 0 | 0 | 1
Not completed — Ongoing Study Period | 2 | 4 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo | Total
Number analyzed (Participants) | 25 | 25 | 24 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 25 | 21 | 68
  >=65 years | 3 | 0 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.3 (15.06) | 42.8 (12.16) | 46.2 (12.82) | 45.4 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 18 | 54
  Male | 8 | 6 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 13 | 27
  Not Hispanic or Latino | 16 | 20 | 11 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 4
  Asian | 2 | 3 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 2 | 12
  White | 17 | 13 | 13 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in CLASI Activity Score at Week 16
Description: The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) is a validated clinical tool designed to assess skin involvement in cutaneous lupus erythematosus (CLE).
  It separately scores:
  * Disease activity (e.g., erythema, scale, mucous membrane involvement, alopecia)
  * Damage (e.g., dyspigmentation, scarring)
  CLASI enables classification of disease severity:
  Mild: Activity score 0-9 Moderate: 10-20 Severe: 21-70
Time Frame: From first dose to Week 16 (approximately 16 weeks)
Population: All Treated Participants in the Placebo Controlled Period with a post baseline measurement in CLASI-A
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 23
Percentage change from baseline | -48.56 (44.684) | -48.93 (33.302) | -27.31 (29.716)

2. Secondary Outcome: Percentage of Participants With an Improvement of ≥ 50% From Baseline in the CLASI-A Score (CLASI-50).
Description: as for outcome 1
Time Frame: From first dose to Week 16 (approximately 16 weeks)
Population: All Treated Participants in the Placebo Controlled Period with a post baseline measurement in CLASI-A
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 23
Percentage of participants | 60.0 | 54.2 | 21.7

3. Secondary Outcome: Percentage of Participants Who Have Disease Improvement as Defined by a Reduction in CLASI-A of ≥ 4 Points From Baseline.
Description: as for outcome 1
Time Frame: From first dose to Week 16 (approximately 16 weeks)
Population: All Treated Participants in the Placebo Controlled Period with a post baseline measurement in CLASI-A
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 23
Percentage of participants | 60.0 | 66.7 | 39.1

4. Secondary Outcome: Mean Change From Baseline in CLASI-A Score.
Description: as for outcome 1
Time Frame: From first dose to Week 16 (approximately 16 weeks)
Population: All Treated Participants in the Placebo Controlled Period with a post baseline measurement in CLASI-A
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 23
Score on a Scale | -9.8 (12.69) | -7.5 (5.92) | -4.3 (5.54)

5. Secondary Outcome: Percentage of Participants Who Have a Complete Response (CR) on CLASI-A Defined as a Score of "0".
Description: The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) is a validated clinical tool designed to assess skin involvement in cutaneous lupus erythematosus (CLE).
  It separately scores:
  * Disease activity (e.g., erythema, scale, mucous membrane involvement, alopecia)
  * Damage (e.g., dyspigmentation, scarring)
  CLASI enables classification of disease severity:
  Mild: Activity score 0-9 Moderate: 10-20 Severe: 21-70
  Complete Response (CR) on CLASI-A defined as a score of "0".
Time Frame: From first dose to Week 16 (approximately 16 weeks)
Population: All Treated Participants in the Placebo Controlled Period with a post baseline measurement in CLASI-A
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 23
Percentage of Participants | 12.0 | 4.2 | 0

6. Secondary Outcome: Number of Participants With Safety Related Events in the Placebo Controlled Period
Description: Number of participants with safety related events in the placebo controlled period
Time Frame: From signing informed consent to end of safety follow up period (Approximately 60 weeks)
Population: All Treated Population in the Placebo Controlled Period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 24
Participants
  TEAE | 17 | 19 | 12
  Treatment-related TEAEs | 11 | 11 | 3
  Serious TEAE | 2 | 2 | 1
  Treatment related Serious TEAE | 1 | 1 | 0

7. Secondary Outcome: Number of Participants With Safety Related Events in the Active Treatment Period
Description: Number of participants with safety related events in the active treatment period
Time Frame: From signing informed consent to end of safety follow up period (Approximately 60 weeks)
Population: All Treated Population in the active treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Active-Treatment Period: Treatment 1 | Active-Treatment Period: Treatment 2
Number analyzed (Participants) | 16 | 20 | 9 | 9
Participants
  TEAEs | 11 | 10 | 5 | 6
  Treatment related TEAEs | 5 | 5 | 2 | 2
  Serious TEAEs | 1 | 0 | 0 | 1
  Treatment related serious TEAE | 1 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in the Placebo Controlled Period
Description: Number of participants with clinically significant laboratory abnormalities in the placebo controlled period
Time Frame: From signing informed consent to end of safety follow up period (Approximately 60 weeks)
Population: All Treated Population in the Placebo Controlled Period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 24
Participants
  Creatinine Kinase ≥ 2.5x ULN: number analyzed (Participants) | 24 | 23 | 22
  Creatinine Kinase ≥ 2.5x ULN | 1 | 1 | 2
  Hemoglobin < 9 g/dL (90g/L): number analyzed (Participants) | 24 | 23 | 22
  Hemoglobin < 9 g/dL (90g/L) | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in the Active Treatment Period
Description: Number of participants with clinically significant laboratory abnormalities in the active treatment period
Time Frame: From signing informed consent to end of safety follow up period (Approximately 60 weeks)
Population: All Treated Population in the active treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Active-Treatment Period: Treatment 1 | Active-Treatment Period: Treatment 2
Number analyzed (Participants) | 16 | 20 | 9 | 9
Participants
  ALT > 3xULN: number analyzed (Participants) | 16 | 19 | 9 | 9
  ALT > 3xULN | 0 | 0 | 1 | 0
  AST > 3xULN: number analyzed (Participants) | 16 | 19 | 9 | 9
  AST > 3xULN | 0 | 0 | 1 | 0
  Creatinine Kinase ≥ 2.5x ULN: number analyzed (Participants) | 16 | 19 | 9 | 9
  Creatinine Kinase ≥ 2.5x ULN | 3 | 1 | 2 | 1
  Hemoglobin < 9 g/dL (90g/L): number analyzed (Participants) | 16 | 19 | 9 | 9
  Hemoglobin < 9 g/dL (90g/L) | 1 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities in the Placebo Controlled Period
Description: Number of participants with clinically significant vital sign abnormalities in the placebo controlled period
Time Frame: From signing informed consent to end of safety follow up period (Approximately 60 weeks)
Population: All Treated Population in the Placebo Controlled Period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 24
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities in the Active Treatment Period
Description: Number of participants with clinically significant vital sign abnormalities in the active treatment period
Time Frame: From signing informed consent to end of safety follow up period (Approximately 60 weeks)
Population: All Treated Population in the active treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Active-Treatment Period: Treatment 1 | Active-Treatment Period: Treatment 2
Number analyzed (Participants) | 16 | 20 | 9 | 9
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant ECG Abnormalities in the Placebo Controlled Period
Description: Number of participants with clinically significant ECG abnormalities in the placebo controlled period
Time Frame: From signing informed consent to end of active treatment period (Approximately 56 weeks)
Population: All Treated Population in the Placebo Controlled Period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Placebo-Controlled Period: Placebo
Number analyzed (Participants) | 25 | 24 | 24
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant ECG Abnormalities in the Active Treatment Period
Description: Number of participants with clinically significant ECG abnormalities in the active treatment period
Time Frame: From signing informed consent to end of active treatment period (Approximately 56 weeks)
Population: All Treated Population in the active treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Period: Treatment 1 | Placebo-Controlled Period: Treatment 2 | Active-Treatment Period: Treatment 1 | Active-Treatment Period: Treatment 2
Number analyzed (Participants) | 16 | 20 | 9 | 9
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs/SAEs are collected from the time of signing the consent until post treatment follow up period of 28 days, approximately 13 months.
Description: The number at Risk for All-Cause Mortality represents all treated participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Placebo-Controlled Period - DEUC 3 mg BID: Deucravactinib 3mg in the Placebo controlled period
- Placebo-Controlled Period - DEUC 6 mg BID: Deucravactinib 6 mg in the Placebo controlled period
- Placebo-Controlled Period - Placebo BID: Placebo in the Placebo controlled period
- Active Treatment Period - DEUC 3 mg BID: Deucravactinib 3mg in the Placebo controlled period and Deucravactinib 3mg in the Active Treatment Period
- Active Treatment Period - DEUC 6 mg BID: Deucravactinib 6mg in the Placebo controlled period and Deucravactinib 6mg in the Active Treatment Period
- Active Treatment Period - Placebo-DEUC 3 mg BID: Placebo in the Placebo controlled period and Deucravactinib 3mg in the Active Treatment Period
- Active Treatment Period - Placebo-DEUC 6 mg BID: Placebo in the Placebo controlled period and Deucravactinib 6mg in the Active Treatment Period
Arm/Group | Placebo-Controlled Period - DEUC 3 mg BID | Placebo-Controlled Period - DEUC 6 mg BID | Placebo-Controlled Period - Placebo BID | Active Treatment Period - DEUC 3 mg BID | Active Treatment Period - DEUC 6 mg BID | Active Treatment Period - Placebo-DEUC 3 mg BID | Active Treatment Period - Placebo-DEUC 6 mg BID
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/24 | 0/16 | 0/20 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/25 | 2/24 | 1/24 | 1/16 | 0/20 | 0/9 | 1/9
Other Adverse Events (participants affected / at risk) | 15/25 | 15/24 | 8/24 | 11/16 | 10/20 | 5/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Period - DEUC 3 mg BID (N=25) | Placebo-Controlled Period - DEUC 6 mg BID (N=24) | Placebo-Controlled Period - Placebo BID (N=24) | Active Treatment Period - DEUC 3 mg BID (N=16) | Active Treatment Period - DEUC 6 mg BID (N=20) | Active Treatment Period - Placebo-DEUC 3 mg BID (N=9) | Active Treatment Period - Placebo-DEUC 6 mg BID (N=9)
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion induced incomplete (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo-Controlled Period - DEUC 3 mg BID (N=25) | Placebo-Controlled Period - DEUC 6 mg BID (N=24) | Placebo-Controlled Period - Placebo BID (N=24) | Active Treatment Period - DEUC 3 mg BID (N=16) | Active Treatment Period - DEUC 6 mg BID (N=20) | Active Treatment Period - Placebo-DEUC 3 mg BID (N=9) | Active Treatment Period - Placebo-DEUC 6 mg BID (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 5 | 1 | 2 | 0
Folliculitis (Infections and infestations) | 2 | 2 | 0 | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 1 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 2 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0/9 | 1/4 | 1/6 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Erythrasma (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pustule (Infections and infestations) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Schistosomiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Nerve degeneration (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1/9 | 0/4 | 0/6 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0/9 | 1/4 | 1/6 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0/9 | 1/4 | 0/6 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0/9 | 0/4 | 1/6 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT04857034/Prot_SAP_000.pdf